CLINICAL TRIAL: NCT06094114
Title: Evaluation of Atrio-ventricular Synchronous Pacing Rate During Exercise Test in Patients With a VDD Leadless Pacing System (Micra AV)
Brief Title: Evaluation of VDD Leadless Pacing System During Exercise
Status: Completed | Type: Observational
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Collaborators: Medtronics, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: s65477
Record Dates: First submitted 2022-11-14; First posted 2023-10-23 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2022-11

CONDITIONS: Bradycardia; Pacemaker DDD
Keywords: leadless pacemaker; Micra
MeSH Terms: conditions — Bradycardia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Patients with Micra Av: Only patients who were previously implanted with a Micra MC1AVR01 can be enrolled in the study. Patients need to be able to perform an exercise test. All subjects provide signed and dated consent that he/she is willing and able to comply with the protocol.
  Interventions: Device: pacemaker follow-up

INTERVENTIONS:
Device: pacemaker follow-up — Performance of an exercise test in patients previously implanted with Micra AV
  Other Names: Micra AV

SUMMARY:
The study is a non-randomized, active prospective observational study permitting to report the behavior of Micra AV pacemaker during an exercise.

Only patients who were previously implanted with a Micra MC1AVR01 can be enrolled in the study. Exercise test is part of the standard clinical care practice for this patients population during the first year follow-up.

DETAILED DESCRIPTION:
The purpose of this observational study is to obtain additional data on behavior and safety of the Micra MC1AVR01 during exercise:

1. Characterize the atrial detection rate/A4 amplitude by a ventricular Micra AV (Micra MC1AVR01) at rest and during exercise
2. Characterize the AV synchrony percentage provided by the Micra AV during exercise.
3. Confirm the safety of the Micra AV during exercise

Only patients who were previously implanted with a Micra MC1AVR01 can be enrolled in the study. All subjects provide signed and dated consent that he/she is willing and able to comply with the protocol.

Retrospective patients enrollment is allowed to facilitate a more rapid performance assessment in patients previously implanted with a Micra AV for whom an exercise test has already been performed.

Exercise test The Micra AV permits AV synchronous pacing mode up to a maximal sinus rate of 115/min. Exercise test will therefore be performed up to a maximal heart rate of 115/min. The test will be stopped by the patient (depending on his/her ability/symptoms such as: fatigue, dyspnea, leg pain,..) or by the cardiologist if a maximal heart rate of 115 beats per minute is reached.

ELIGIBILITY:
Inclusion Criteria:

* Patients previously implanted with a Micra MC1AVR01
* Signed and dated consent (patient confirms that he/she is willing and able to comply with the protocol)
* Patient is physically able to perform an exercise test (cycle test).

Retrospective patients enrolment is allowed to facilitate a more rapid performance assessment in patients previously implanted with a Micra AV for whom an exercise test has already been performed.

Co-enrolment in the Micra AV post-approvals study is allowed.

Exclusion Criteria:

- Frail patient unable to perform an exercise test (cycle test).

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients previously implanted with Micra AV
Sampling Method: Non-Probability Sample
Enrollment: 42 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Characterize the atrial detection rate/A4 amplitude by a ventricular Micra AV (Micra MC1AVR01) at rest and during exercise | Exercise test is performed during the first year following the Micra implantation
  Characterize the atrial detection rate/A4 amplitude by a ventricular Micra AV (Micra MC1AVR01) at rest and during exercise
Characterize the AV synchrony percentage provided by the Micra AV during exercise. | Exercise test is performed during the first year following the Micra implantation
  Characterize the AV synchrony percentage provided by the Micra AV during exercise.
Confirm the safety of the Micra AV during exercise | Exercise test is performed during the first year following the Micra implantation
  Confirm the safety of the Micra AV during exercise confirmed by the absence of (1) pauses exceeding 2 paced cardiac cycles and (2) oversensing induced tachyarrhythmia exceeding 130 bpm.

CONTACTS AND LOCATIONS:
Overall Officials: Christophe Garweg, MD,PHD, Principal Investigator — University Hospitals of Leuven, cardiovascular department
Locations (1):
- University Hospitals of Leuven, Leuven, Belgium

IPD SHARING:
Plan to Share IPD: No